CLINICAL TRIAL: NCT00368641
Title: Treatment-Resistant Heart Failure (HF) and Peritoneal Ultrafiltration (PUF): A Randomized Prospective Trial of Standard Care Versus Standard Care With Peritoneal Ultrafiltration in Patients With Treatment-Resistant Severe Heart Failure
Brief Title: Heart Failure and Peritoneal Ultrafiltration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Former Sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25885
Record Dates: First submitted 2006-08-23; First posted 2006-08-25 (Estimated); Results first posted 2009-06-17 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Icodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): peritoneal dialysis
  Interventions: Drug: Extraneal
- Standard of Care (No Intervention)

INTERVENTIONS:
Drug: Extraneal — Periotneal Dialysis
  Arms: Intervention

SUMMARY:
The objective of the study is to determine if the addition of peritoneal ultrafiltration to standard therapy in treatment-resistant severe heart failure patients will improve fluid balance and functional capacity such that they will spend less time in the hospital and have an improved ambulatory quality of life in comparison to patients who remain on standard therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults with congestive heart failure (CHF) who remain fluid overloaded despite standard treatment.

Exclusion Criteria:

* Patients who have reversible CHF or have diseases or conditions that would contraindicate the use of peritoneal dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - San Jose, California
  - Torrance, California
  - Denver, Colorado
  - Evanston, Illinois
  - Winston-Salem, North Carolina
- Melbourne, Victoria, Australia
- Belgium (3):
  - Leuven
  - Liège
  - Roeselare
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 sites were active to enroll subjects from March 2, 2007 through February 29, 2008
Pre-assignment Details: Subjects were required to meet all inclusion and no exclusion criteria for study participation
Groups:
- Intervention Group: Addition of peritoneal ultrafiltration
- Standard Therapy: Standard therapy for CHF
Period: Overall Study
Arm/Group | Intervention Group | Standard Therapy
Started | 6 | 6
Completed | 0 (study was terminated prior to completion of treatment period) | 0 (study was terminated prior to completion of treatment period)
Not Completed | 6 | 6
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Sponsor decision to terminate study | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Standard Therapy | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.8 (4.1) | 70.7 (13.1) | 74.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4.0
  Canada | 3 | 3 | 6.0
  Belgium | 1 | 1 | 2.0

OUTCOME MEASURES:

1. Primary Outcome: All-cause Hospitalization (Unadjusted)
Description: All-cause hospitalization was defined as (1) hospitalization for any cause of any duration or (2)any ER visit or any clinic visit specifically for congestive heart failure requiring intravenous administration of an inotrope, vasodilator or diuretic.
Time Frame: 6 to 24 months
Population: intent to treat population
Measure: Mean (95% Confidence Interval); unit: hospitalizations per year
Arm/Group | Intervention Group | Standard Therapy
Number analyzed (Participants) | 6 | 6
hospitalizations per year | 5.33 [3.13 to 9.05] | 1.69 [0.95 to 2.99]

ADVERSE EVENTS:
Arm/Group | Intervention Group | Standard Therapy
Serious Adverse Events (participants affected / at risk) | 6 | 4
Other Adverse Events (participants affected / at risk) | 6 | 6
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Intervention Group | Standard Therapy
pneumonia (Infections and infestations) | 0/6 (0) | 1/6 (1)
fluid overload (Metabolism and nutrition disorders) | 0/6 (0) | 1/6 (1)
chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/6 (0) | 1/6 (1)
cellulitis (Infections and infestations) | 0/6 (0) | 1/6 (1)
hyperkalaemia (Metabolism and nutrition disorders) | 0/6 (0) | 1/6 (1)
renal failure (Renal and urinary disorders) | 0/6 (0) | 1/6 (1)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/6 (1)
cardiac failure congestive (Cardiac disorders) | 2/6 (2) | 1/6 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/6 (1) | 0/6 (0)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/6 (1) | 0/6 (0)
diabetic gastroparesis (Gastrointestinal disorders) | 1/6 (1) | 0/6 (0)
catheter related complication (General disorders) | 1/5 (1) | 0/0 (0)
fungal peritonitis (Infections and infestations) | 1/5 (1) | 0/0 (0)
renal failure acute (Renal and urinary disorders) | 1/6 (1) | 0/6 (0)
shock (Vascular disorders) | 1/6 (1) | 0/6 (0)
jaundice (Hepatobiliary disorders) | 1/6 (1) | 0/6 (0)
peritonitis bacterial (Infections and infestations) | 1/5 (1) | 0/0 (0)
cardiac arrest (Cardiac disorders) | 1/6 (1) | 0/6 (0)
peritonitis (Gastrointestinal disorders) | 1/5 (1) | 0/0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Intervention Group | Standard Therapy
anaemia (Blood and lymphatic system disorders) | 1/6 (1) | 1/6 (1)
cardiac failure congestive (Cardiac disorders) | 3/6 (3) | 3/6 (3)
nausea (Gastrointestinal disorders) | 2/6 (2) | 1/6 (1)
constipation (Gastrointestinal disorders) | 1/6 (1) | 0/6 (0)
gastrooesophageal reflux disease (Gastrointestinal disorders) | 1/6 (1) | 0/6 (0)
megacolon (Gastrointestinal disorders) | 1/6 (1) | 0/6 (0)
vomiting (Gastrointestinal disorders) | 0/6 (0) | 1/6 (1)
catheter site pain (General disorders) | 3/6 (3) | 0/0 (0)
asthenia (General disorders) | 0/6 (0) | 1/6 (1)
catheter site erythema (General disorders) | 1/6 (1) | 0/0 (0)
chest pain (General disorders) | 0/6 (0) | 1/6 (1)
fatigue (General disorders) | 0/6 (0) | 1/6 (1)
local swelling (General disorders) | 1/6 (1) | 0/6 (0)
oedema (General disorders) | 0/6 (0) | 1/6 (1)
oedema peripheral (General disorders) | 0/6 (0) | 1/6 (1)
pyrexia (General disorders) | 1/6 (1) | 0/6 (0)
catheter site infection (Infections and infestations) | 2/6 (2) | 0/0 (0)
bronchitis (Infections and infestations) | 0/6 (0) | 1/6 (1)
bursitis infective (Infections and infestations) | 0/6 (0) | 1/6 (1)
escherichia urinary tract infection (Infections and infestations) | 1/6 (1) | 0/6 (0)
nasopharyngitis (Infections and infestations) | 0/6 (0) | 1/6 (1)
respiratory tract infection (Infections and infestations) | 0/6 (0) | 1/6 (1)
upper respiratory tract infection (Infections and infestations) | 1/6 (1) | 0/6 (0)
contusion (Injury, poisoning and procedural complications) | 0/6 (0) | 1/6 (1)
excoriation (Injury, poisoning and procedural complications) | 0/6 (0) | 1/6 (1)
fall (Injury, poisoning and procedural complications) | 1/6 (1) | 0/6 (0)
post procedural nausea (Injury, poisoning and procedural complications) | 1/6 (1) | 0/0 (0)
blood glucose increased (Investigations) | 0/6 (0) | 1/6 (1)
international normalized ratio decreased (Investigations) | 1/6 (1) | 0/6 (0)
hypokalaemia (Metabolism and nutrition disorders) | 2/6 (2) | 1/6 (1)
fluid overload (Metabolism and nutrition disorders) | 1/6 (1) | 0/6 (0)
anorexia (Metabolism and nutrition disorders) | 1/6 (1) | 0/6 (0)
gout (Metabolism and nutrition disorders) | 0/6 (0) | 1/6 (1)
hyperglycaemia (Metabolism and nutrition disorders) | 1/6 (1) | 0/6 (0)
hyperlipidaemia (Metabolism and nutrition disorders) | 0/6 (0) | 1/6 (1)
hyperuricaemia (Metabolism and nutrition disorders) | 0/6 (0) | 1/6 (1)
hypocalcaemia (Metabolism and nutrition disorders) | 1/6 (1) | 0/6 (0)
hypocholesterolaemia (Metabolism and nutrition disorders) | 1/6 (1) | 0/6 (0)
hypoglycaemia (Metabolism and nutrition disorders) | 1/6 (1) | 0/6 (0)
hyponatraemia (Metabolism and nutrition disorders) | 0/6 (0) | 1/6 (1)
lactic acidosis (Metabolism and nutrition disorders) | 1/6 (1) | 0/6 (0)
bursitis (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/6 (1)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/6 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/6 (1)
dizziness (Nervous system disorders) | 0/6 (0) | 2/6 (2)
ageusia (Nervous system disorders) | 0/6 (0) | 1/6 (1)
myoclonus (Nervous system disorders) | 1/6 (1) | 0/6 (0)
tremor (Nervous system disorders) | 0/6 (0) | 1/6 (1)
confusional state (Psychiatric disorders) | 1/6 (1) | 2/6 (2)
agitation (Psychiatric disorders) | 1/6 (1) | 0/6 (0)
anxiety (Psychiatric disorders) | 1/6 (1) | 0/6 (0)
micturition urgency (Renal and urinary disorders) | 0/6 (0) | 1/6 (1)
renal disorder (Renal and urinary disorders) | 0/6 (0) | 1/6 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/6 (1) | 1/6 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1/6 (1) | 1/6 (1)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1/6 (1) | 1/6 (1)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/6 (1) | 0/6 (0)
productive cough (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/6 (1)
sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/6 (1)
sneezing (Respiratory, thoracic and mediastinal disorders) | 1/6 (1) | 0/6 (0)
haemmorrhage (Vascular disorders) | 0/6 (0) | 1/6 (1)
cardiac failure (Cardiac disorders) | 0/6 (0) | 1/6 (1)

LIMITATIONS AND CAVEATS:
The number of subjects enrolled & duration of therapy were insufficient to complete the planned efficacy analyses & to draw any conclusion regarding all-cause hospitalization rates in both intervention and standard therapy arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No